CLINICAL TRIAL: NCT06749171
Title: Comparative Analysis of Coronary Revascularization Approaches Within Gender and Sex Aspects
Brief Title: Coronary Revascularization Outcomes Within Necessary Sex and Gender Aspects
Acronym: CROWN-SAGA
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Institution "Federal Center for Cardiovascular Surgery named after S.G. Sukh (Other)
Responsible Party: Principal Investigator, Lilothia Sofia Harishevna, MD, Cardiovascular Surgeon, Federal State Budgetary Institution "Federal Center for Cardiovascular Surgery named after S.G. Sukh
Other Study IDs: CROWN-SAGA
Record Dates: First submitted 2024-12-09; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease; Coronary Artery Bypass Grafting
Keywords: coronary artery bypass grafting; revascularization; OPCAB; ONCAB; NTA; MICSCAB; multiple arterial grafting; sequential grafts; composite grafts; cardiac surgery; women; sex; gender
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coitus | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women: Women undergoing CABG
  Interventions: Procedure: coronary artery bypass grafting
- Men: Men undergoing CABG
  Interventions: Procedure: coronary artery bypass grafting

INTERVENTIONS:
Procedure: coronary artery bypass grafting — ONCAB (on-pump coronary artery bypass grafting), OPCAB (off-pump coronary artery bypass grafting), NTA (no-touch aorta technique), MICSCAB (minimally invasive multiple coronary artery bypass grafting)

SUMMARY:
The aim of this observational single-centre study is the optimization of coronary artery bypass grafting (CABG) tactics considering gender and sex approach on the basis of complex comparative evaluation of surgical revascularization techniques. Patients enrolled in the study are divided into groups based on sex, as well as into stratum of surgery techniques.

Objectives of the study are:

1. To evaluate the preoperative profile of women and men referred for CABG.
2. To give a comparative assessment of CABG outcomes in the short-term and long-term postoperative period in patients of both sexes.
3. To carry out the comparative analysis of short-term and long-term outcomes of different CABG techniques for each sex.
4. To analyse the causes and identify predictors of complications and mortality after CABG in the female and male cohort.
5. To determine an optimal selection strategy of surgical revascularization technique for patients of different sexes based on the conducted comparative gender-sex analysis of modern coronary surgery techniques.

DETAILED DESCRIPTION:
This retrospective-prospective single-centre study aims to conduct an in-depth comparative analysis of the impact of preoperative profile and range of surgical techniques in coronary artery bypass grafting (CABG) surgery on short-term and long-term outcomes in women and men.

The study included a sample of 400 patients (200 women and 200 men) who underwent CABG between January 2016 and July 2023. Patients enrolled in the study were divided into groups based on sex with the following propensity score matching (PSM) analysis, as well as into stratum of surgery techniques - ONCAB (on-pump coronary artery bypass grafting), OPCAB (off-pump coronary artery bypass grafting), NTA (no-touch aorta technique), MICSCAB (minimally invasive multiple coronary artery bypass grafting). Furthermore, the impact of multiple arterial grafting (MAG), total arterial revascularization (TAR), composite and sequential grafting on outcomes was analyzed for each sex.

Included patients were evaluated for 112 various parameters of preoperative profile, intraoperative characteristics, in-hospital and long-term postoperative data. Perioperative data was obtained from the centre's digital medical information system. Long-term data was gathered from the regional state health information system by tracking patients' chronology of outpatient visits and complaints, subsequent hospital admissions, clinical and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* patients with multivessel coronary artery disease requiring CABG;
* age ≥ 18 years;
* patients residing in the Perm region.

Exclusion Criteria:

* single-vessel CABG;
* redo CABG;
* concomitant coronary artery disease and caroid artery disease and/or valvular disease and/or rhythm disorders requiring surgical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were sampled from a cohort of 7945 CABG patients in accordance with the eligibility criteria and time period, followed by use of random number generating method to enrol 200 females and 200 males.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
MACCE | from date of hospital discharge until the date of first documented major adverse cardiac and cerebrovascular event, through study completion, up to an average of 30 months
  major adverse cardiac and cerebrovascular events - composite of all-cause mortality, myocardial infarction (MI), stroke or transient ischaemic attack (TIA) and repeat revascularization

SECONDARY OUTCOMES:
Death | from date of hospital discharge until the date of death from any cause, through study completion, up to an average of 30 months
  all-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Centre for Cardiovascular Surgery n.a. S.G. Sukhanov, Perm, Perm Kray, Russia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lilothia S.H. Timeline of scientific knowledge in the field of coronary artery bypass surgery focusing in the gender and sex perspective. Complex Issues of Cardiovascular Diseases. 2024;13(2): 196-202. DOI: 10.17802/2306-1278-202413-2-196-202
- [Background] Lilothia S. H. Gender inequality and cardiovascular diseases. Russian Journal of Cardiology. 2024;29(6):5873. doi: 10.15829/1560-4071-2024-5873. EDN LPEYQM